CLINICAL TRIAL: NCT02535754
Title: Interventions to Increase Workplace Wellness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H10-01079
Record Dates: First submitted 2015-08-24; First posted 2015-08-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ALIVE (Experimental): Email program N=170
  Interventions: Behavioral: ALIVE
- CCS BCY (Experimental): Comprehensive program N=285
  Interventions: Behavioral: CCS BCY
- ALIVE + CCS BCY (Experimental): Email + comprehensive program N=225
  Interventions: Behavioral: ALIVE + CCS BCY

INTERVENTIONS:
Behavioral: ALIVE — The company assigned to this condition offered employees participation in the ALIVE program. This program was validated in a previous worksite-based randomized controlled trial (RCT). A baseline assessment includes questions asking about: presence of children at home, habits related to cooking and eating out, physical activity preferences, stage of readiness of change, and perceived barriers to achieving heath behavior goals. This information provides the basis for immediate feedback and individually-tailored messages that include goal-setting and tips to achieve these goals, interactive features, and health information. Biweekly messages are sent for a total of 48 weeks. Outcome data were based on all individuals who completed the baseline assessment.
  Arms: ALIVE
Behavioral: CCS BCY — The company assigned to this condition participated in a comprehensive year-long workplace wellness program intervention focusing on nutrition, weight control, and physical activity, led by the CCS BCY. The program was modeled after a previous successful CCS BCY tobacco control worksite program. This program stresses the importance of developing social and environmental supports at the worksite to promote behavior change . Such supports could include food availability (e.g., cafeteria and vending machine selections), the built environment (e.g., availability of bike racks); social environment (e.g., group lunchtime walking clubs), and health communications (e.g., company newsletters). Outcome data were based on all individuals who completed the baseline assessment.
  Arms: CCS BCY
Behavioral: ALIVE + CCS BCY — The company assigned to this condition received both the ALIVE and CCS BCY programs. Employees were encouraged to take part in both ALIVE and company initiatives, but participation in these activities was based on individual preference. Outcome data were based on all individuals who completed the baseline assessment.
  Arms: ALIVE + CCS BCY

SUMMARY:
Behaviour changes such as improving nutrition, increasing physical activity, and decreasing obesity are linked with lower mortality and morbidity and fewer cancers. Health promotion programs in the workplace are a promising way to reach a large segment of the population. This project evaluated the efficacy of three approaches - all of which were based on previous research and programs with demonstrated positive benefits - on cancer-related outcomes (healthy eating, physical activity, normal body weight) and work-related outcomes (absenteeism, presenteeism).

DETAILED DESCRIPTION:
The project evaluated the efficacy of three health promotion interventions on cancer- and work-related outcomes. Three worksites in British Columbia were randomly assigned to one of three conditions: (1) an empirically-validated intervention directed at individual behavior change using personally-tailored messages delivered by email (ALIVE) ; (2) a comprehensive approach building on social and institutional support developed by the Canadian Cancer Society British Columbia Yukon and previously used for worksite tobacco control (CCS BCY) and (3) an intervention including both of these approaches (CCS BCY + ALIVE). The primary outcome was change in fruit and vegetable consumption from baseline to 16 months, as an indicator of healthy diet. Change in weight, physical activity, and work productivity were secondary outcomes. The investigators also conducted focus groups to assess participant perspectives on the programs which comprise another secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Employee of the company
* English speaking with reading level at Flesch-Kincaid 8.5 grade level
* Ability to provide access to individual work email address

Exclusion Criteria:

* Non-English speaking without reading level at Flesch-Kincaid 8.5 grade level
* Inability to provide access to individual work email address

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 682 (Actual)
Dates: Start 2010-04; Primary Completion 2013-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in number of fruit and vegetable servings per day | 16 months
  Self-reported number of fruit and vegetable servings at baseline and 16 months

SECONDARY OUTCOMES:
Absenteeism (days) | 16 months
  Self-reported absenteeism at baseline and 16 months
Change in body weight (lbs) | 16 months
  Self-reported height and weight at baseline and 16 months
Physical activity efficacy (minutes) | 16 months
  Self-reported efficacy for physical activity at baseline and 16 months
Participant perspectives on the program (theme) | 16 months
  Focus groups identified participant responses to the program including strengths and weaknesses.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn C Gotay, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada